CLINICAL TRIAL: NCT03281304
Title: A PHASE 3B/4, MULTI-CENTER, DOUBLE-BLIND, RANDOMIZED, PARALLEL GROUP STUDY OF TOFACITINIB (CP-690,550) IN SUBJECTS WITH ULCERATIVE COLITIS IN STABLE REMISSION
Brief Title: A Study of Tofacitinib in Patients With Ulcerative Colitis in Stable Remission
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study terminated early due to business reasons, with the study already meeting its primary objective. The decision to terminate the trial was not based on any safety and/or efficacy concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921288; RIVETING STUDY (Other: Alias Study Number); 2017-002274-39 (EudraCT Number)
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Results first posted 2021-04-15 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-02

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis; inflammatory bowel disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CP-690,550 5 mg (Experimental): CP-690,550 5 mg tablet by mouth twice a day (BID)
  Interventions: Drug: CP-690,500 5 mg
- CP-690,550 10 mg (Experimental): CP-690,550 10 mg BID
  Interventions: Drug: CP-690,550 10 mg

INTERVENTIONS:
Drug: CP-690,500 5 mg — CP-690,550 5 mg tablet BID
  Arms: CP-690,550 5 mg
Drug: CP-690,550 10 mg — CP-690,550 10 mg tablet BID
  Arms: CP-690,550 10 mg

SUMMARY:
This study is a follow up study for subjects with Ulcerative Colitis (UC) in stable remission designed to evaluate flexible dosing of CP-690,550.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in Study A3921139 receiving CP-690,550 10 mg BID for at least 2 years consecutively.
* In stable remission on CP-690,550 10 mg BID
* Agree to use highly effective contraception
* Negative pregnancy test
* Comply with visits, treatments, lab tests, diary and other study procedures
* Signed and dated informed consent document.

Exclusion Criteria:

* Subjects who were initially assigned to tofacitinib 10 mg BID at baseline of Study A3921139 whose tofacitinib dose was reduced to 5 mg BID due to safety or efficacy.
* Presence of indeterminate colitis, microscopic colitis, ischemic colitis, infectious colitis or findings suggestive of Crohn's disease
* Likely to require surgery for ulcerative colitis during study
* Expected to receive any prohibited medication
* Expected to receive live or attenuated virus vaccination during study
* Women who are pregnant or breastfeeding or planning to become pregnant during the study
* Evidence of colonic malignancy or any dysplasia
* Acute or chronic medical or psychiatric condition that may increase risk of participation
* Investigator site staff member
* Subjects likely to be uncooperative or unable to comply with study procedures
* Participation in other studies involving investigational drugs during study
* Subjects with any of the following risk factors for pulmonary embolism at baseline as defined by EMA's PRAC:

  * has heart failure;
  * has inherited coagulation disorders;
  * has had venous thromboembolism, either deep venous thrombosis or pulmonary embolism;
  * is taking combined hormonal contraceptives or hormone replacement therapy;
  * has malignancy (association is strongest with cancers other than non-melanoma skin cancers);
  * is undergoing major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2022-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (80):
- United States (24):
  - Surgicare of Mobile, Mobile, Alabama
  - Alabama Medical Group, P.C., Mobile, Alabama
  - Clinical Applications Laboratories, Inc., San Diego, California
  - Bristol Hospital, Bristol, Connecticut
  - Connecticut Clinical Research Institute, Bristol, Connecticut
  - Central Connecticut Endoscopy Center, Plainville, Connecticut
  - Advanced Medical Research Center, Port Orange, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - Chevy Chase Endoscopy Center, Chevy Chase, Maryland
  - MGG Group Co., Inc., Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Eastside Endoscopy Center, Macomb, Michigan
  - Clinical Research Institute of Michigan, LLC, Troy, Michigan
  - NYU Langone Long Island Clinical Research Associates, Lake Success, New York
  - Columbia University Irving Medical Center, New York, New York
  - Columbia University Medical Center Research Pharmacy/ Milstein Hospital, New York, New York
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Memorial Hermann Hospital, Houston, Texas
  - The University of Texas Health Science Center at Houston (UTHealth)- McGovern Medical School, Houston, Texas
  - Christus Trinity Mother Frances Endoscopy Center, Tyler, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Alpine Medical Group, Salt Lake City, Utah
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
- UZ Leuven (University Hospital Leuven), Campus Gasthuisberg, Leuven, Belgium
- Canada (2):
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Royal University Hospital, Saskatoon, Saskatchewan
- Nemocnice Strakonice a.s., Strakonice, Czechia
- France (2):
  - CHU Hotel Dieu, Nantes
  - CHU de Bordeaux Hopital Haut Leveque, Pessac
- Universitaetsklinikum Schleswig-Holstein, Kiel, Germany
- Hungary (3):
  - Szent Janos Korhaz és Eszak-budai Egyesitett Korhazak, Budapest
  - Pannonia Maganorvosi Centrum Kft., Budapest
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaz Endoszkopos Laboratorium, Gyula
- Università "Magna Graecia" di Catanzaro, Catanzaro, CZ, Italy
- Japan (14):
  - Aichi Medical University Hospital, Nagakute, Aichi-ken
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Hokkaido P.W.F.A.C Sapporo-Kosei General Hospital, Sapporo, Hokkaido
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki-shi, Osaka
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Tokyo Medical And Dental University Hospital, Faculty of Medicine, Bunkyo-ku, Tokyo
  - Tokai University Hachioji Hospital, Hachiōji, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - Showa University Hospital, Shinagawa-ku, Tokyo
  - Toho University Sakura Medical Center, Chiba
  - Hiroshima University Hospital, Hiroshima
  - Osaka Metropolitan University Hospital, Osaka
  - Keio University Hospital, Tokyo
- Academic Medical Centre, Amsterdam, Netherlands
- New Zealand (3):
  - North Shore Hospital (Waitemata District Health Board), Takapuna, Auckland
  - Christchurch Hospital (Canterbury District Health Board), Christchurch
  - Southern District Health Board, Dunedin
- Poland (2):
  - Endoskopia Sp. z o.o., Sopot
  - Lexmedica, Wroclaw
- Russia (3):
  - Federal State Budgetary Institution "State Scientific Centre of Coloproctology, Moscow
  - LLC Novosibirskiy Gastrocenter, Novosibirsk
  - Federal State Budgetary Scientific Institution "Scientific Research Institute of Physiology, Novosibirsk
- Serbia (5):
  - Clinical Centre of Serbia, Clinic for Gastroenterology and Hepatology, Belgrade
  - Clinical Hospital Centre Zvezdara, Belgrade
  - Military Medical Academy, Clinic for Gastroenterology and Hepatology, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - General Hospital "Djordje Joanovic", Zrenjanin
- Slovakia (3):
  - Medak s.r.o., Bratislava
  - KM Management spol. s.r.o., Nitra
  - Gastro I., s.r.o., Gastroenterologicka ambulancia, Prešov
- South Africa (5):
  - Kingsbury Hospital, Claremont, CAPE TOWN
  - Wits Clinical Research (WCR) Bara Site, Chris Hani Baragwanath Academic Hospital, Soweto, Johannesburg, Gauteng
  - Chris Hani Baragwanath Academic Hospital, Soweto, Johannesburg
  - Endocare Research Centre, Paarl, Western Cape
  - Panorama Mediclinic, Panorama, Western Cape
- South Korea (3):
  - Hanyang University Guri Hospital, Gyeonggi-do
  - Kyung Hee University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Hospital Clinic de Barcelona, Barcelona, Spain
- Ukraine (4):
  - Regional Municipal Non-Profit Enterprise "Chernivtsi Regional Clinical Hospital" Surgery Departm, Chernivtsi
  - Kyiv Municipal Clinical Hospital #18, Kyiv
  - MI Uzhgorod Regional Hospital, Uzhhorod
  - Vinnytsia Regional Clinical Hospital for War Veterans, Therapeutics Dept. No. 2, Vinnytsia
- University Hospitals Bristol NHS Foundation Trust, Bristol, AVON, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Torres J, D'Haens GR, Regueiro M, Santana G, Panes J, Vermeire S, Gardiner S, Kulisek N, Modesto I, Su C, Lawendy N, Mundayat R, Paulissen J, Dubinsky MC. Potential predictors of efficacy outcomes following tofacitinib dose reduction in patients with ulcerative colitis in stable remission: a post hoc analysis of outcomes from the RIVETING study. Therap Adv Gastroenterol. 2025 Feb 27;18:17562848251318849. doi: 10.1177/17562848251318849. eCollection 2025. PMID 40028509
- [Derived] Panes J, D'Haens GR, Sands BE, Ng SC, Lawendy N, Kulisek N, Guo X, Wu J, Vranic I, Panaccione R, Vermeire S. Analysis of tofacitinib safety in ulcerative colitis from the completed global clinical developmental program up to 9.2 years of drug exposure. United European Gastroenterol J. 2024 Jul;12(6):793-801. doi: 10.1002/ueg2.12584. Epub 2024 May 22. PMID 38778549
- [Derived] Rubin DT, Torres J, Regueiro M, Reinisch W, Prideaux L, Kotze PG, Tan FH, Gardiner S, Mundayat R, Cadatal MJ, Ng SC. Association Between Smoking Status and the Efficacy and Safety of Tofacitinib in Patients with Ulcerative Colitis. Crohns Colitis 360. 2024 Jan 20;6(1):otae004. doi: 10.1093/crocol/otae004. eCollection 2024 Jan. PMID 38425446
- [Derived] Sandborn WJ, D'Haens GR, Sands BE, Panaccione R, Ng SC, Lawendy N, Kulisek N, Modesto I, Guo X, Mundayat R, Su C, Vranic I, Panes J. Tofacitinib for the Treatment of Ulcerative Colitis: An Integrated Summary of up to 7.8 Years of Safety Data from the Global Clinical Programme. J Crohns Colitis. 2023 Apr 3;17(3):338-351. doi: 10.1093/ecco-jcc/jjac141. PMID 36124702
- [Derived] Winthrop KL, Vermeire S, Long MD, Panes J, Ng SC, Kulisek N, Mundayat R, Lawendy N, Vranic I, Modesto I, Su C, Melmed GY. Long-term Risk of Herpes Zoster Infection in Patients With Ulcerative Colitis Receiving Tofacitinib. Inflamm Bowel Dis. 2023 Jan 5;29(1):85-96. doi: 10.1093/ibd/izac063. PMID 35648151
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921288

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled participants from A3921139 (NCT01470612) who were on tofacitinib 10 milligram (mg) twice daily (BID) for at least 2 consecutive years, who were in stable remission for at least 6 months prior to baseline of A3921288 and who were not receiving any corticosteroid treatment to treat their ulcerative colitis (UC) for at least 4 weeks prior to enrollment.
Pre-assignment Details: The Baseline visit of this study was the last visit in study A3921139. All procedures done at the last visit in A3921139 for participants enrolled into this study were used as the Baseline data for this study.
Groups:
- Tofacitinib 5 mg BID: Participants received tofacitinib 5 mg tablet with one tablet of matching placebo, orally, twice daily up to 42 months. Participants were followed up to 4 weeks after the last dose.
- Tofacitinib 10 mg BID: Participants received tofacitinib 10 mg tablets (2 tablets of 5 mg), orally, twice daily up to 42 months. Participants were followed up to 4 weeks after the last dose.
Period: Treatment Phase (up to 42 Months)
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Started | 70 | 70
Completed | 36 | 27
Not Completed | 34 | 43
Not completed — Adverse Event | 10 | 10
Not completed — Lack of Efficacy | 3 | 2
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 5 | 12
Not completed — Death | 0 | 1
Not completed — Study terminated by sponsor | 15 | 16
Not completed — Other | 0 | 2
Period: Follow-up Phase (up to 4 Weeks)
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Started | 63 (Participants could be followed up even if they did not complete treatment.) | 57 (Participants could be followed up even if they did not complete treatment.)
Completed | 61 | 56
Not Completed | 2 | 1
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who were randomized and received at least 1 dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 63 | 122
  >=65 years | 11 | 7 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 44 | 48 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 68 | 67 | 135
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 14 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 50 | 50 | 100
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Remission Based on Modified Mayo Score at Month 6
Description: Remission as per modified mayo score was defined as an endoscopic subscore of 0 or 1, stool frequency subscore of 0 or 1, and rectal bleeding subscore of 0 at Month 6. Modified mayo score consisted of 3 components: stool frequency subscore, rectal bleeding subscore and endoscopic subscore: higher scores for each score = more severe disease. These scores were summed up to give a total modified mayo score range of 0 to 9; where higher scores indicating more severe disease.
Time Frame: Month 6
Population: Full analysis set included all participants who were randomized and received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 70 | 70
Participants | 54 | 63
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Adjusted (weighted) difference and its 95% CI based on normal approximation for the difference in binomial proportions; Test type: Other; Adjusted (weighted) difference = 12.9, 95% CI 2-sided [0.5 to 25.0]

2. Secondary Outcome: Time to Loss of Remission Based on Modified Mayo Score Using Kaplan-Meier Method
Description: Time to loss of remission(flare): time from first drug administration until time of meeting loss of remission criteria based on modified mayo score. Loss of remission: meeting at least (>=)1 criteria: increase from Baseline in rectal bleeding subscore by >=1 point and increase in endoscopic subscore by >=1 point; increase from Baseline in rectal bleeding subscore by >=2 points and endoscopic subscore >0; increase in stool frequency subscore by >=2 points and increase in endoscopic subscore by >=1 point; increase in endoscopic subscore by >=2 points. Modified mayo score included 3 components: stool frequency, rectal bleeding and endoscopic subscores: Modified mayo score included 3 components: stool frequency, rectal bleeding and endoscopic subscores, each subscore graded from 0 to 3 with higher scores for each score=more severe disease. All scores summed up to give total modified mayo score range from 0 to 9; higher scores=more severe disease.
Time Frame: Up to Month 42
Population: Full analysis set included all participants who were randomized and received at least 1 dose of investigational product.
Measure: Median (Full Range); unit: Days
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 70 | 70
Days | NA [29 to 1268] — Median was not estimated due to insufficient number of participants with the event. | 1270 [28 to 1270]

3. Secondary Outcome: Number of Participants With Remission Based on Modified Partial Mayo Score at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39 and 42
Description: Remission as per modified partial mayo score was defined as stool frequency subscore of 0 or 1, and rectal bleeding sub score of 0 at the specified time points. Modified partial mayo scores consisted of 2 components: stool frequency and rectal bleeding: each subscore graded from 0 to 3 with higher scores for each score = more severe disease. These scores were summed up to give a total modified partial mayo score range of 0 to 6; where higher scores indicating more severe disease.
Time Frame: Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39 and 42
Population: Full analysis set included all participants who were randomized and received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 70 | 70
Participants
  Month 1 | 62 | 64
  Month 3 | 57 | 65
  Month 6 | 57 | 67
  Month 9 | 52 | 66
  Month 12 | 50 | 61
  Month 15 | 48 | 58
  Month 18 | 45 | 55
  Month 21 | 46 | 51
  Month 24 | 47 | 51
  Month 27 | 43 | 49
  Month 30 | 44 | 46
  Month 33 | 42 | 43
  Month 36 | 42 | 44
  Month 39 | 40 | 37
  Month 42 | 26 | 29
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 1: Adjusted (weighted) difference and its 95% CI based on normal approximation for the difference in binomial proportions; Test type: Other; Adjusted (weighted) difference = 2.9, 95% CI 2-sided [-7.5 to 13.4]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 3: Adjusted (weighted) difference and its 95% CI based on normal approximation for the difference in binomial proportions; Test type: Other; Adjusted (weighted) difference = 11.4, 95% CI 2-sided [0.1 to 22.8]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 6: Adjusted (weighted) difference and its 95% CI based on normal approximation for the difference in binomial proportions; Test type: Other; Adjusted (weighted) difference = 14.3, 95% CI 2-sided [2.9 to 25.2]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 9: Adjusted (weighted) difference and its 95% CI based on normal approximation for the difference in binomial proportions; Test type: Other; Adjusted (weighted) difference = 20.0, 95% CI 2-sided [8.0 to 31.8]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 12: Adjusted (weighted) difference and its 95% CI based on normal approximation for the difference in binomial proportions; Test type: Other; Adjusted (weighted) difference = 15.7, 95% CI 2-sided [2.2 to 28.7]
Statistical Analysis 6: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 15: Adjusted (weighted) difference and its 95% CI based on normal approximation for the difference in binomial proportions; Test type: Other; Adjusted (weighted) difference = 14.3, 95% CI 2-sided [0.0 to 27.9]
Statistical Analysis 7: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 18: Adjusted (weighted) difference and its 95% CI based on normal approximation for the difference in binomial proportions; Test type: Other; Adjusted (weighted) difference = 14.3, 95% CI 2-sided [-0.7 to 28.5]
Statistical Analysis 8: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 21: Adjusted (weighted) difference and its 95% CI based on normal approximation for the difference in binomial proportions; Test type: Other; Adjusted (weighted) difference = 7.1, 95% CI 2-sided [-8.0 to 21.9]
Statistical Analysis 9: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 24: Adjusted (weighted) difference and its 95% CI based on normal approximation for the difference in binomial proportions; Test type: Other; Adjusted (weighted) difference = 5.7, 95% CI 2-sided [-9.3 to 20.4]
Statistical Analysis 10: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 27: Adjusted (weighted) difference and its 95% CI based on normal approximation for the difference in binomial proportions; Test type: Other; Adjusted (weighted) difference = 8.6, 95% CI 2-sided [-7.0 to 23.6]
Statistical Analysis 11: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 30: Adjusted (weighted) difference and its 95% CI based on normal approximation for the difference in binomial proportions; Test type: Other; Adjusted (weighted) difference = 2.9, 95% CI 2-sided [-12.8 to 18.3]
Statistical Analysis 12: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 33: Adjusted (weighted) difference and its 95% CI based on normal approximation for the difference in binomial proportions; Test type: Other; Adjusted (weighted) difference = 1.4, 95% CI 2-sided [-14.4 to 17.2]
Statistical Analysis 13: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 36: Adjusted (weighted) difference and its 95% CI based on normal approximation for the difference in binomial proportions; Test type: Other; Adjusted (weighted) difference = 2.9, 95% CI 2-sided [-13.0 to 18.5]
Statistical Analysis 14: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 39: Adjusted (weighted) difference and its 95% CI based on normal approximation for the difference in binomial proportions; Test type: Other; Adjusted (weighted) difference = -4.3, 95% CI 2-sided [-20.2 to 11.9]
Statistical Analysis 15: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 42: Adjusted (weighted) difference and its 95% CI based on normal approximation for the difference in binomial proportions; Test type: Other; Adjusted (weighted) difference = 4.3, 95% CI 2-sided [-11.7 to 19.9]

4. Secondary Outcome: Number of Participants With Remission Based on Total Mayo Score at Months 6, 18, 30 and 42
Description: Remission as per total mayo score was defined by a total mayo score of 2 points or lower, with no individual subscore exceeding 1 point and a rectal bleeding subscore of 0. Mayo score is an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of flexible sigmoidoscopy and physician global assessment (PGA), each subscore graded from 0 to 3 with higher scores indicating more severe disease. PGA included 3 criteria: participant's recollection of abdominal discomfort, general sense of wellbeing and other observations such as physical findings and performance status. Individual subscores were summed up to give a total mayo score range of 0 to 12, where higher scores indicating more severe disease.
Time Frame: Months 6, 18, 30 and 42
Population: Full analysis set included all participants who were randomized and received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 70 | 70
Participants
  Month 6 | 53 | 61
  Month 18 | 33 | 47
  Month 30 | 35 | 44
  Month 42 | 22 | 24
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 3]; Test type: Other; Adjusted (weighted) difference = 11.4, 95% CI 2-sided [-1.5 to 24.1]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 7]; Test type: Other; Adjusted (weighted) difference = 20.0, 95% CI 2-sided [3.6 to 35.0]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 11]; Test type: Other; Adjusted (weighted) difference = 12.9, 95% CI 2-sided [-3.5 to 28.3]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 15]; Test type: Other; Adjusted (weighted) difference = 2.9, 95% CI 2-sided [-12.5 to 18.0]

5. Secondary Outcome: Number of Participants With Remission Based on Partial Mayo Score at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39 and 42
Description: Remission as per partial mayo score was defined as partial mayo score of 2 points or lower, with no individual subscore exceeding 1 point and a rectal bleeding subscore of 0. Partial mayo score was an instrument designed to measure disease activity of UC without endoscopy. It consisted of 3 subscores: stool frequency, rectal bleeding and PGA with each subscore graded from 0 to 3 with higher scores indicating more severe disease. PGA included 3 criteria: participant's recollection of abdominal discomfort, general sense of wellbeing and other observations such as physical findings and performance status. Individual subscores were summed up to give a total partial mayo score range from 0 (normal or inactive disease) to 9 (severe disease) with higher scores indicating more severe disease.
Time Frame: Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39 and 42
Population: Full analysis set included all participants who were randomized and received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 70 | 70
Participants
  Month 1 | 62 | 64
  Month 3 | 57 | 65
  Month 6 | 56 | 66
  Month 9 | 52 | 66
  Month 12 | 50 | 61
  Month 15 | 48 | 58
  Month 18 | 44 | 55
  Month 21 | 46 | 50
  Month 24 | 46 | 51
  Month 27 | 42 | 49
  Month 30 | 43 | 46
  Month 33 | 42 | 43
  Month 36 | 42 | 44
  Month 39 | 39 | 37
  Month 42 | 26 | 28
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 1]; Test type: Other; Adjusted (weighted) difference = 2.9, 95% CI 2-sided [-7.5 to 13.4]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 2]; Test type: Other; Adjusted (weighted) difference = 11.4, 95% CI 2-sided [0.1 to 22.8]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 3]; Test type: Other; Adjusted (weighted) difference = 14.3, 95% CI 2-sided [2.4 to 25.6]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 4]; Test type: Other; Adjusted (weighted) difference = 20.0, 95% CI 2-sided [8.0 to 31.8]
Statistical Analysis 5: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 5]; Test type: Other; Adjusted (weighted) difference = 15.7, 95% CI 2-sided [2.2 to 28.7]
Statistical Analysis 6: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 6]; Test type: Other; Adjusted (weighted) difference = 14.3, 95% CI 2-sided [0.0 to 27.9]
Statistical Analysis 7: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 7]; Test type: Other; Adjusted (weighted) difference = 15.7, 95% CI 2-sided [0.7 to 29.9]
Statistical Analysis 8: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 8]; Test type: Other; Adjusted (weighted) difference = 5.7, 95% CI 2-sided [-9.5 to 20.6]
Statistical Analysis 9: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 9]; Test type: Other; Adjusted (weighted) difference = 7.1, 95% CI 2-sided [-8.0 to 21.9]
Statistical Analysis 10: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 10]; Test type: Other; Adjusted (weighted) difference = 10.0, 95% CI 2-sided [-5.7 to 25.1]
Statistical Analysis 11: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 11]; Test type: Other; Adjusted (weighted) difference = 4.3, 95% CI 2-sided [-11.4 to 19.7]
Statistical Analysis 12: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 12]; Test type: Other; Adjusted (weighted) difference = 1.4, 95% CI 2-sided [-14.4 to 17.2]
Statistical Analysis 13: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 13]; Test type: Other; Adjusted (weighted) difference = 2.9, 95% CI 2-sided [-13.0 to 18.5]
Statistical Analysis 14: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 14]; Test type: Other; Adjusted (weighted) difference = -2.9, 95% CI 2-sided [-18.8 to 13.3]
Statistical Analysis 15: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 15]; Test type: Other; Adjusted (weighted) difference = 2.9, 95% CI 2-sided [-13.0 to 18.5]

6. Secondary Outcome: Number of Participants With Remission Based on Modified Mayo Score at Months 18, 30 and 42
Description: Remission as per modified mayo score was defined as an endoscopic subscore of 0 or 1, stool frequency subscore of 0 or 1, and rectal bleeding subscore of 0. Modified mayo score consisted of 3 components: stool frequency subscore, rectal bleeding subscore and endoscopic subscore: higher scores for each score = more severe disease. These scores were summed up to give a total modified mayo score range of 0 to 9; where higher scores indicating more severe disease.
Time Frame: Months 18, 30 and 42
Population: Full analysis set included all participants who were randomized and received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 70 | 70
Participants
  Month 18 | 37 | 48
  Month 30 | 35 | 44
  Month 42 | 23 | 24
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 7]; Test type: Other; Adjusted (weighted) difference = 15.7, 95% CI 2-sided [-0.4 to 30.8]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 11]; Test type: Other; Adjusted (weighted) difference = 12.9, 95% CI 2-sided [-3.5 to 28.3]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 15]; Test type: Other; Adjusted (weighted) difference = 1.4, 95% CI 2-sided [-14.0 to 16.7]

7. Secondary Outcome: Change From Baseline in Modified Mayo Score at Month 6
Description: Modified mayo score is an instrument designed to measure disease activity of UC. Modified mayo scores consisted of 3 subscores: stool frequency, rectal bleeding and endoscopic subscore, each subscore graded from 0 to 3 with higher scores indicating more severe disease. These individual scores were summed up to give a total modified mayo score range of 0 to 9, where higher scores indicated more severe disease.
Time Frame: Baseline, Month 6
Population: Full analysis set included all participants who were randomized and received at least 1 dose of investigational product. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 67 | 68
Units on a scale | 0.6 (0.2) | 0.3 (0.2)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Test type: Other; Mean Difference = -0.3, 95% CI 2-sided [-0.8 to 0.1]

8. Secondary Outcome: Change From Baseline in Modified Mayo Score at Months 18, 30 and 42
Description: as for outcome 7
Time Frame: Baseline, Months 18, 30 and 42
Population: Full analysis set included all participants who were randomized and received at least 1 dose of investigational product. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and 'Number Analyzed' = participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 48 | 57
Units on a scale
  Change at Month 18 | 0.5 (1.3) | 0.3 (1.5)
  Change at Month 30: number analyzed (Participants) | 44 | 45
  Change at Month 30 | 0.3 (1.2) | 0.1 (0.9)
  Change at Month 42: number analyzed (Participants) | 40 | 34
  Change at Month 42 | 0.3 (0.9) | 0.2 (1.1)

9. Secondary Outcome: Change From Baseline in Modified Partial Mayo Score at Months 1, 3 and 6
Description: Modified partial mayo scores consisted of 2 subscores: stool frequency and rectal bleeding with each subscore graded from 0 to 3 with higher scores indicating more severe disease. Individual subscores were summed up to give a total Modified partial mayo score ranges from 0 (normal or inactive disease) to 6 (severe disease) with higher scores indicating more severe disease.
Time Frame: Baseline, Months 1, 3 and 6
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 67 | 69
Units on a scale
  Change at Month 1: number analyzed (Participants) | 67 | 66
  Change at Month 1 | 0.1 (0.1) | 0.2 (0.1)
  Change at Month 3: number analyzed (Participants) | 64 | 68
  Change at Month 3 | 0.2 (0.1) | 0.1 (0.1)
  Change at Month 6: number analyzed (Participants) | 60 | 69
  Change at Month 6 | 0.1 (0.1) | 0.2 (0.1)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 1; Test type: Other; Least Squares (LS) Mean Difference = 0.1, 95% CI 2-sided [-0.1 to 0.3]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 3; Test type: Other; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.2]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 6; Test type: Other; LS Mean Difference = 0.0, 95% CI 2-sided [-0.2 to 0.3]

10. Secondary Outcome: Change From Baseline in Modified Partial Mayo Score at Months 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39 and 42
Description: Modified partial mayo scores consisted of 2 subscores: stool frequency and rectal bleeding with each subscore graded from 0 to 3 with higher scores indicating more severe disease. Individual subscores were summed up to give a total modified partial mayo score range from 0 (normal or inactive disease) to 6 (severe disease) with higher scores indicating more severe disease.
Time Frame: Baseline, Months 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39 and 42
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 53 | 67
Units on a scale
  Change at Month 9 | 0.1 (0.7) | 0.1 (0.6)
  Change at Month 12: number analyzed (Participants) | 51 | 63
  Change at Month 12 | 0.1 (0.5) | 0.1 (0.7)
  Change at Month 15: number analyzed (Participants) | 51 | 57
  Change at Month 15 | 0.2 (0.8) | 0.1 (0.6)
  Change at Month 18: number analyzed (Participants) | 47 | 56
  Change at Month 18 | 0.1 (0.6) | 0.1 (0.8)
  Change at Month 21: number analyzed (Participants) | 48 | 54
  Change at Month 21 | 0.1 (0.5) | 0.2 (1.1)
  Change at Month 24: number analyzed (Participants) | 47 | 50
  Change at Month 24 | 0.0 (0.5) | 0.0 (0.6)
  Change at Month 27: number analyzed (Participants) | 45 | 48
  Change at Month 27 | 0.1 (0.5) | 0.1 (0.7)
  Change at Month 30: number analyzed (Participants) | 45 | 45
  Change at Month 30 | 0.1 (0.7) | 0.0 (0.6)
  Change at Month 33: number analyzed (Participants) | 42 | 41
  Change at Month 33 | 0.0 (0.4) | 0.2 (0.7)
  Change at Month 36: number analyzed (Participants) | 43 | 41
  Change at Month 36 | 0.0 (0.5) | 0.0 (0.5)
  Change at Month 39: number analyzed (Participants) | 40 | 34
  Change at Month 39 | 0.0 (0.5) | 0.0 (0.5)
  Change at Month 42: number analyzed (Participants) | 26 | 26
  Change at Month 42 | 0.1 (0.4) | 0.1 (0.7)

11. Secondary Outcome: Change From Baseline in Total Mayo Score at Month 6
Description: Mayo score is an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of flexible sigmoidoscopy and PGA, each sub score graded from 0 to 3 with higher scores indicating more severe disease. PGA included 3 criteria: participant's recollection of abdominal discomfort, general sense of wellbeing and other observations such as physical findings and performance status. Individual subscores were summed up to give a total mayo score range of 0 to 12, where higher scores indicating more severe disease.
Time Frame: Baseline, Month 6
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 67 | 68
Units on a scale | 0.9 (0.2) | 0.4 (0.3)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Test type: Other; LS Mean Difference = -0.6, 95% CI 2-sided [-1.2 to 0.1]

12. Secondary Outcome: Change From Baseline in Total Mayo Score at Months 18, 30 and 42
Description: as for outcome 11
Time Frame: Baseline, Months 18, 30 and 42
Population: Full analysis set included all participants who were randomized and received at least 1 dose of investigational product. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed"= participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 48 | 57
Units on a scale
  Change at Month 18 | 0.7 (1.7) | 0.4 (1.9)
  Change at Month 30: number analyzed (Participants) | 44 | 45
  Change at Month 30 | 0.4 (1.4) | 0.1 (1.2)
  Change at Month 42: number analyzed (Participants) | 40 | 34
  Change at Month 42 | 0.4 (1.2) | 0.2 (1.4)

13. Secondary Outcome: Change From Baseline in Partial Mayo Score at Months 1, 3 and 6
Description: Partial mayo score was an instrument designed to measure disease activity of UC without endoscopy. It consisted of 3 subscores: stool frequency, rectal bleeding and PGA with each subscore graded from 0 to 3 with higher scores indicating more severe disease. PGA included 3 criteria: participant's recollection of abdominal discomfort, general sense of wellbeing and other observations such as physical findings and performance status. Individual subscores were summed up to give a total partial mayo score range from 0 (normal or inactive disease) to 9 (severe disease) with higher scores indicating more severe disease.
Time Frame: Baseline, Months 1, 3 and 6
Population: Full analysis set included all participants who were randomized and received at least 1 dose of investigational product. Here, 'Number Analyzed' = participants evaluable for this outcome measure at specified time points.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 70 | 70
Units on a scale
  Change at Month 1: number analyzed (Participants) | 67 | 66
  Change at Month 1 | 0.2 (0.1) | 0.2 (0.1)
  Change at Month 3: number analyzed (Participants) | 64 | 68
  Change at Month 3 | 0.3 (0.1) | 0.2 (0.1)
  Change at Month 6: number analyzed (Participants) | 60 | 69
  Change at Month 6 | 0.3 (0.1) | 0.3 (0.1)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 1; Test type: Other; LS Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.3]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 3; Test type: Other; LS Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.2]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; Month 6; Test type: Other; LS Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.3]

14. Secondary Outcome: Change From Baseline in Partial Mayo Score at Months 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39 and 42
Description: Partial mayo score was an instrument designed to measure disease activity of UC without endoscopy. It consisted of 3 subscores: stool frequency, rectal bleeding and PGA with each subscore graded from 0 to 3 with higher scores indicating more severe disease. PGA included 3 criteria: participant's recollection of abdominal discomfort, general sense of wellbeing and other observations such as physical findings and performance status. Individual subscores were summed up to give a total partial mayo score ranges from 0 (normal or inactive disease) to 9 (severe disease) with higher scores indicating more severe disease.
Time Frame: Baseline, Months 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39 and 42
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 53 | 67
Units on a scale
  Change at Month 9 | 0.2 (0.8) | 0.2 (0.9)
  Change at Month 12: number analyzed (Participants) | 51 | 63
  Change at Month 12 | 0.1 (0.7) | 0.2 (0.9)
  Change at Month 15: number analyzed (Participants) | 51 | 57
  Change at Month 15 | 0.3 (1.2) | 0.1 (0.8)
  Change at Month 18: number analyzed (Participants) | 47 | 56
  Change at Month 18 | 0.2 (0.8) | 0.2 (1.2)
  Change at Month 21: number analyzed (Participants) | 48 | 54
  Change at Month 21 | 0.1 (0.7) | 0.4 (1.7)
  Change at Month 24: number analyzed (Participants) | 46 | 50
  Change at Month 24 | 0.1 (0.6) | 0.0 (0.8)
  Change at Month 27: number analyzed (Participants) | 44 | 48
  Change at Month 27 | 0.1 (0.6) | 0.1 (0.9)
  Change at Month 30: number analyzed (Participants) | 45 | 45
  Change at Month 30 | 0.2 (0.8) | 0.1 (0.8)
  Change at Month 33: number analyzed (Participants) | 42 | 41
  Change at Month 33 | 0.0 (0.5) | 0.2 (1.0)
  Change at Month 36: number analyzed (Participants) | 43 | 41
  Change at Month 36 | 0.0 (0.6) | -0.1 (0.6)
  Change at Month 39: number analyzed (Participants) | 39 | 34
  Change at Month 39 | 0.1 (0.6) | -0.1 (0.6)
  Change at Month 42: number analyzed (Participants) | 26 | 25
  Change at Month 42 | 0.1 (0.5) | 0.2 (1.1)

15. Secondary Outcome: Number of Participants With Mucosal Healing at Months 6, 18, 30 and 42
Description: Mucosal healing in participants was defined as the mayo endoscopic subscore of 0 or 1. The Mayo endoscopic subscore consisted of the findings of centrally read flexible sigmoidoscopy, graded from 0 to 3 with higher scores indicated more severe disease.
Time Frame: Months 6, 18, 30 and 42
Population: Full analysis set included all participants who were randomized and received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 70 | 70
Participants
  Month 6 | 56 | 64
  Month 18 | 43 | 56
  Month 30 | 38 | 47
  Month 42 | 36 | 36
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 3]; Test type: Other; Adjusted (weighted) difference = 11.4, 95% CI 2-sided [-0.3 to 23.1]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 7]; Test type: Other; Adjusted (weighted) difference = 18.6, 95% CI 2-sided [3.5 to 32.6]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 11]; Test type: Other; Adjusted (weighted) difference = 12.9, 95% CI 2-sided [-3.3 to 28.1]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 15]; Test type: Other; Adjusted (weighted) difference = 0.0, 95% CI 2-sided [-16.1 to 16.1]

16. Secondary Outcome: Number of Participants With Clinical Response Based on Mayo Score at Months 6, 18, 30 and 42
Description: Clinical response was defined as a decrease from baseline in mayo score of at least 3 points and at least 30 percent, with an accompanying decrease in the rectal bleeding subscore of at least 1 point or an absolute rectal bleeding subscore of 0 or 1. Mayo score is an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of flexible sigmoidoscopy and PGA, each sub score graded from 0 to 3 with higher scores indicating more severe disease. PGA included 3 criteria: participant's recollection of abdominal discomfort, general sense of wellbeing and other observations such as physical findings and performance status. Individual subscores were summed up to give a mayo score range of 0 to 12, where higher scores indicating more severe disease.
Time Frame: Months 6, 18, 30 and 42
Population: Full analysis set included all participants who were randomized and received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 70 | 70
Participants
  Month 6 | 59 | 67
  Month 18 | 42 | 50
  Month 30 | 41 | 48
  Month 42 | 26 | 28
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 3]; Test type: Other; Adjusted (weighted) difference = 11.4, 95% CI 2-sided [1.3 to 22.0]
Statistical Analysis 2: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 7]; Test type: Other; Adjusted (weighted) difference = 11.4, 95% CI 2-sided [-4.2 to 26.4]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 11]; Test type: Other; Adjusted (weighted) difference = 10.0, 95% CI 2-sided [-5.8 to 25.2]
Statistical Analysis 4: Comparison: Tofacitinib 5 mg BID vs Tofacitinib 10 mg BID; [analysis description as in outcome 3, analysis 15]; Test type: Other; Adjusted (weighted) difference = 2.9, 95% CI 2-sided [-13.0 to 18.5]

17. Secondary Outcome: Change From Baseline in Fecal Calprotectin at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39 and 42
Description: Change from baseline in fecal calprotectin (in micrograms per gram [mcg/g]) was reported.
Time Frame: Baseline, Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39 and 42
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Micrograms per gram
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 63 | 67
Micrograms per gram
  Change at Month 1: number analyzed (Participants) | 63 | 62
  Change at Month 1 | -137.5 (980.6) | -21.9 (304.7)
  Change at Month 3: number analyzed (Participants) | 57 | 63
  Change at Month 3 | -45.3 (1075.8) | -38.5 (313.6)
  Change at Month 6: number analyzed (Participants) | 52 | 67
  Change at Month 6 | -24.1 (1444.6) | -47.3 (331.4)
  Change at Month 9: number analyzed (Participants) | 48 | 62
  Change at Month 9 | -173.5 (1106.5) | -59.3 (380.8)
  Change at Month 12: number analyzed (Participants) | 46 | 54
  Change at Month 12 | -28.8 (1113.4) | -45.0 (350.7)
  Change at Month 15: number analyzed (Participants) | 45 | 49
  Change at Month 15 | -104.8 (1210.2) | 69.3 (480.5)
  Change at Month 18: number analyzed (Participants) | 39 | 44
  Change at Month 18 | -51.0 (1114.6) | 6.6 (565.4)
  Change at Month 21: number analyzed (Participants) | 43 | 46
  Change at Month 21 | -71.0 (1254.6) | -29.3 (462.7)
  Change at Month 24: number analyzed (Participants) | 41 | 43
  Change at Month 24 | 118.3 (1591.4) | -69.8 (407.0)
  Change at Month 27: number analyzed (Participants) | 38 | 39
  Change at Month 27 | 87.3 (478.8) | -49.1 (366.3)
  Change at Month 30: number analyzed (Participants) | 36 | 40
  Change at Month 30 | -8.5 (458.5) | -8.9 (518.5)
  Change at Month 33: number analyzed (Participants) | 36 | 38
  Change at Month 33 | 84.4 (434.5) | -4.9 (484.8)
  Change at Month 36: number analyzed (Participants) | 38 | 36
  Change at Month 36 | 230.7 (1162.5) | -0.4 (449.4)
  Change at Month 39: number analyzed (Participants) | 28 | 26
  Change at Month 39 | -116.2 (472.8) | -98.3 (532.9)
  Change at Month 42: number analyzed (Participants) | 24 | 23
  Change at Month 42 | -44.7 (278.9) | -101.0 (452.0)

18. Secondary Outcome: Change From Baseline in High Sensitivity C-Reactive Protein (Hs-CRP) Level at Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39 and 42
Description: Change From baseline in hs-CRP level (in milligrams per liter [mg/L]) is reported.
Time Frame: Baseline, Months 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39 and 42
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Milligrams per liter
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 63 | 67
Milligrams per liter
  Change at Month 1 | 1.1 (9.8) | -0.7 (3.4)
  Change at Month 3: number analyzed (Participants) | 56 | 66
  Change at Month 3 | 0.7 (7.9) | -0.2 (3.7)
  Change at Month 6: number analyzed (Participants) | 55 | 66
  Change at Month 6 | 0.9 (5.8) | 0.1 (4.0)
  Change at Month 9: number analyzed (Participants) | 50 | 63
  Change at Month 9 | 0.7 (11.1) | 1.1 (8.4)
  Change at Month 12: number analyzed (Participants) | 48 | 59
  Change at Month 12 | -0.3 (3.5) | -0.2 (2.2)
  Change at Month 15: number analyzed (Participants) | 46 | 51
  Change at Month 15 | -0.7 (3.2) | 0.2 (2.4)
  Change at Month 18: number analyzed (Participants) | 43 | 48
  Change at Month 18 | 1.0 (6.4) | 0.2 (1.9)
  Change at Month 21: number analyzed (Participants) | 44 | 49
  Change at Month 21 | -0.5 (3.3) | -0.1 (1.4)
  Change at Month 24: number analyzed (Participants) | 40 | 43
  Change at Month 24 | -0.6 (3.0) | -0.5 (2.2)
  Change at Month 27: number analyzed (Participants) | 39 | 42
  Change at Month 27 | -0.3 (2.8) | 0.7 (6.1)
  Change at Month 30: number analyzed (Participants) | 39 | 44
  Change at Month 30 | 0.6 (4.1) | -0.3 (1.9)
  Change at Month 33: number analyzed (Participants) | 38 | 39
  Change at Month 33 | 0.1 (2.2) | 0.0 (3.9)
  Change at Month 36: number analyzed (Participants) | 38 | 36
  Change at Month 36 | -0.1 (3.1) | -0.1 (3.9)
  Change at Month 39: number analyzed (Participants) | 37 | 34
  Change at Month 39 | -0.3 (3.5) | 2.8 (8.6)
  Change at Month 42: number analyzed (Participants) | 27 | 25
  Change at Month 42 | 0.6 (3.7) | 5.9 (28.1)

19. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment or worsened during the treatment period relative to the pretreatment state. AEs included both serious and all non-serious adverse events (irrespective of frequency threshold used to report other AEs in safety section).
Time Frame: Baseline up to 43 months
Population: Safety analysis set included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 70 | 70
Participants
  TEAEs | 55 | 58
  SAEs | 7 | 16

20. Secondary Outcome: Number of Participants With Serious Infections
Description: Serious infections were defined as any infections (viral, bacterial, and fungal) requiring parenteral antimicrobial therapy, hospitalization for treatment, or meeting other criteria that require the infection to be classified as serious adverse event. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events.
Time Frame: Baseline up to 43 months
Population: Safety analysis set included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 70 | 70
Participants | 3 | 6

21. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: Abnormality criteria: Hematology: hemoglobin(Hg): <0.8* lower limit of normal (LLN); hematocrit: <0.8*LLN; lymphocytes: <0.8* LLN; lymphocytes/leukocytes: <0.8*LLN; erythrocytes: <0.8*LLN; erythrocytes mean corpuscular volume: <0.9*LLN; erythrocytes mean corpuscular Hg: <0.9*LLN; reticulocytes, reticulocytes/erythrocytes:>1.5* upper limit of normal (ULN); neutrophils, neutrophils/leukocytes: >1.2*ULN; basophils/leukocytes, eosinophils, eosinophils/leukocytes, monocytes/leukocytes: >1.2*ULN; leukocyte esterase: >=1; Clinical chemistry: bicarbonate:<0.9*LLN, bilirubin: >1.5*ULN; indirect bilirubin: >1.5* ULN; aspartate aminotransferase(AT): >3.0*ULN; alanine AT: >3.0*ULN; gamma glutamyl transferase: >3.0* ULN; creatine kinase: >2.0*ULN; potassium: >1.1*ULN; blood urea nitrogen: >1.3*ULN; creatinine: >1.3*ULN; urate: >1.2*ULN; cholesterol: >1.3*ULN; HDL-cholesterol: <0.8* LLN; LDL-cholesterol: >1.2*ULN; triglycerides: >1.3*ULN; glucose: >1.5*ULN; and urine Hg >=1.
Time Frame: Baseline up to 27 months
Population: Safety analysis set included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 70 | 70
Participants | 33 | 51

22. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities Leading to Study Treatment Discontinuation
Description: Laboratory abnormalities leading to study treatment discontinuation: 2 sequential neutrophil counts <750 neutrophils per cubic millimeter (mm^3); 2 sequential lymphocyte counts <500 lymphocytes/mm^3; 2 sequential hemoglobin <8.0 grams per deciliter; 2 sequential platelet counts <75000 platelets/mm^3; 2 sequential AST or ALT elevations >=3*ULN with at least one total bilirubin value >=2*ULN; 2 sequential AST or ALT elevations >=3*ULN accompanied by signs or symptoms consistent with hepatic injury; 2 sequential AST or ALT elevations >=5*ULN; 2 sequential increases in creatinine >50% and >0.5 milligrams per deciliter over A3921139 baseline; 2 sequential CK elevations >10*ULN unless the causality is known not to be medically serious (eg, exercise induced).
Time Frame: Baseline up to 43 months
Population: Safety analysis set included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 70 | 70
Participants | 1 | 1

23. Secondary Outcome: Number of Participants With Vital Sign Abnormalities
Description: Vital signs abnormality criteria included: 1) a) diastolic blood pressure (DBP) of (less than) <50 millimeter of mercury (mmHg), b) change greater than equal to (>=) 20 mmHg increase, c) change >=20 mmHg decrease; 2) a) systolic blood pressure (SBP) of <90 mmHg, b) change >=30 mmHg increase, c) change >=30 mmHg decrease; 3) a) pulse rate value of <40 beats per minute (bpm), b) pulse rate >120 bpm. Only those categories in which at least 1 participant had data were reported.
Time Frame: Baseline up to 43 months
Population: Safety analysis set included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 70 | 70
Participants
  DBP: <50 mmHg | 3 | 0
  DBP: Change >= 20mmHg increase | 9 | 5
  DBP: Change >= 20mmHg decrease | 7 | 7
  SBP: <90mmHg | 2 | 0
  SBP: Change >= 30mmHg increase | 7 | 4
  SBP: Change >= 30mmHg decrease | 6 | 6

24. Secondary Outcome: Number of Participants With Clinically Significant Physical Examinations Abnormalities
Description: Physical examination included assessment of the weight, general appearance, eyes, mouth, lungs, heart, abdomen, musculoskeletal, extremities, skin and lymph nodes. Clinical significance was assessed by the Investigator.
Time Frame: Baseline up to 43 months
Population: Safety analysis set included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 70 | 70
Participants | 28 | 27

25. Secondary Outcome: Number of Participants With Opportunistic Infections, All Malignancy, Gastrointestinal Perforation and Cardiovascular Events Adjudicated by Adjudication Committee
Description: Number of participants with adjudicated opportunistic infections including herpes zoster (non-adjacent or >2 adjacent dermatomes); all malignancies including non-melanoma skin cancer; gastrointestinal perforation and cardiovascular events including pulmonary embolism and cerebrovascular accident, adjudicated by adjudication committee were reported.
Time Frame: Baseline up to 43 months
Population: Safety analysis set included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 70 | 70
Participants
  Opportunistic Infections | 0 | 1
  All Malignancy | 4 | 3
  Gastrointestinal Perforation | 0 | 0
  Cardiovascular Events | 2 | 2

ADVERSE EVENTS:
Time Frame: From baseline up to 4 weeks after last dose (maximum up to 43 months)
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis set included all participants who received at least 1 dose of investigational product.
Groups:
- Tofacitinib 10 mg BID: Participants received tofacitinib 10 mg tablets (2 tablets of 5 mg), orally, twice daily up to 42 months. Participants were followed-up to 4 weeks after the last dose.
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
All-Cause Mortality (participants affected / at risk) | 0/70 | 1/70
Serious Adverse Events (participants affected / at risk) | 7/70 | 16/70
Other Adverse Events (participants affected / at risk) | 47/70 | 47/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 5 mg BID (N=70) | Tofacitinib 10 mg BID (N=70)
Angina pectoris (Cardiac disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Breast disorder (Reproductive system and breast disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Colon dysplasia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 2
COVID-19 pneumonia (Infections and infestations) | 0 | 2
Herpes zoster oticus (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 5 mg BID (N=70) | Tofacitinib 10 mg BID (N=70)
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Colitis ulcerative (Gastrointestinal disorders) | 16 | 14
Large intestine polyp (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 3 | 3
Oedema peripheral (General disorders) | 2 | 2
Bronchitis (Infections and infestations) | 1 | 5
Herpes zoster (Infections and infestations) | 2 | 5
Influenza (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 7 | 8
Oral herpes (Infections and infestations) | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 3
Blood creatine phosphokinase increased (Investigations) | 2 | 5
Faecal calprotectin increased (Investigations) | 1 | 3
Lymphocyte count decreased (Investigations) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Headache (Nervous system disorders) | 4 | 3
Hypertension (Vascular disorders) | 4 | 5
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Lymphopenia (Blood and lymphatic system disorders) | 2 | 5
Atrial fibrillation (Cardiac disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 0
Chest pain (General disorders) | 2 | 0
Fatigue (General disorders) | 2 | 0
Pyrexia (General disorders) | 5 | 2
COVID-19 (Infections and infestations) | 2 | 0
Clostridium difficile infection (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
SARS-CoV-2 test positive (Investigations) | 2 | 7
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT03281304/Prot_001.pdf
  • Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT03281304/SAP_000.pdf